CLINICAL TRIAL: NCT04389242
Title: An Evidence-based Program Evaluation of the Effectiveness of Internet-based Cognitive Behavioral Preventive Intervention in Reducing Psychological Distress for Chinese University Students in Hong Kong
Brief Title: Online Cognitive Behavioral Intervention Program for Hong Kong University Students
Acronym: REST Online
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Stockholm University (Other); Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Jiayan Pan, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12606118
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Psychological Distress

STUDY DESIGN:
Intervention Model Description: Online Cognitive Behavioral Therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- web-based cognitive behavioral intervention (Experimental): The web-based program is consisted of 8 online modules, forum, internal messaging, reminder, online assessment and online booking. Each online module contains mood check, animation briefing and debriefing, case demonstration videos, session review and exercise.
  Blended mode is adopted to deliver service, which includes the online program, one face-to-face session and one telephone follow-up with a certified CBT therapist.
  Interventions: Other: REST Online（Reduce Stress Tour Online）
- app-based cognitive behavioral intervention (Experimental): Application-based cognitive behavioral intervention program The App-based program is consisted of 8 online modules, forum, internal messaging, reminder, online assessment and online booking. Each online module contains mood check, animation briefing and debriefing, case demonstration videos, session review and exercise.
  Blended mode is adopted to deliver service, which includes the online program, one face-to-face session and one telephone follow-up with a certified CBT therapist.
  Interventions: Other: REST Online（Reduce Stress Tour Online）
- Wait-list control group (Other): No intervention will be provided when the experimental groups are receiving services, but the access to the App-based program will be delivered to the wait-list control group after the two experimental groups complete the service.
  Interventions: Other: REST Online（Reduce Stress Tour Online）

INTERVENTIONS:
Other: REST Online（Reduce Stress Tour Online） — Different cognitive behavioral skills are introduced and practiced in a 8 weekly online program, which includes animation briefing and debriefing, case demonstration video, exercise, forum, internal messaging, online assessment and reminder. One face-to-face session and one telephone follow-up provided by an experienced CBT therapist are also provided to clients.

SUMMARY:
Brief summary:

The objective of this study is to develop an internet-based cognitive behavioral intervention program (including an online platform and a smartphone application) for Chinese university students in Hong Kong, and examine its effectiveness in reducing psychological distress, anxiety/depression symptoms, and improving emotions and automatic thoughts. The 3-month maintenance effect will also be tested.

DETAILED DESCRIPTION:
Previous research has provided evidence for the effectiveness of internet-based cognitive behavioral intervention in improving mental health, but most studies were done in Western countries. This study is intended to design a culturally appropriate online program especially for Chinese university students in Hong Kong. The program will include 8 weekly sessions and one face-to-face session and one telephone follow-up with a with certified CBT therapist. The effects on psychological distress, anxiety/depression, emotions, and automatic thoughts will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Chinese nationality
* Has mild to moderate level of psychological distress
* Receive no face-to-face counselling since program commencement

Exclusion Criteria:

* Has low/high level of psychological distress
* Has one or more psychosis
* Has suicidal risk in the past 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire-12 (GHQ-12) | 3 months
  12 item rating scale for psychological distress.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | 3 months
  21-item rating scale for depressive symptoms.
Beck Anxiety Inventory (BAI) | 3 months
  21-item rating scale for cognitive and somatic symptoms of anxiety.
Chinese Automatic Thoughts Questionnaire (CATQ) | 3 months
  20-item rating scale for automatic thoughts.
Chinese Affect Scale (CAS) | 3 months
  20-item rating scale for affect state of Chinese-speaking people.
Electronic Learning Satisfaction Scale (ELSS) (administered at post-test only)) | 2 months
  17-item rating scale for satisfaction toward electronic learning

CONTACTS AND LOCATIONS:
Overall Officials: Jiayan Pan, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Jiayan Pan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No